CLINICAL TRIAL: NCT04042545
Title: SAFETY AND EFFICACY OF PPP001-kit FOR THE UNCONTROLLED PAIN RELIEF IN PATIENTS WITH ADVANCED CANCER: A RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, PARALLEL GROUP STUDY
Brief Title: Safety and Efficacy of Inhaled Cannabis For the Uncontrolled Pain Relief in Patients With Advanced Cancer
Acronym: PLENITUDE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tetra Bio-Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PPP001-Ph2-02
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-02

CONDITIONS: Cancer Pain; Quality of Life; Pain, Acute; Cannabis Use
MeSH Terms: conditions — Cancer Pain; Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- inhaled THC/CBD (PPP001) (Experimental): PPP001 (cannabis dosing capsule with THC/CBD) inhalation with a device
  Interventions: Drug: PPP001
- Placebo (Placebo Comparator): Placebo inhalation with a device
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PPP001 — 1 cannabis dosing capsule inhaled 3 times a day with a vaporizer device
  Other Names: QIXLEEF
  Arms: inhaled THC/CBD (PPP001)
Drug: Placebo — 1 placebo dosing capsule inhaled 3 times a day with a vaporizer device
  Arms: Placebo

SUMMARY:
This phase 2 multicenter clinical trial assess the safety and efficacy of inhaled PPP001 to relieve the pain in 78 advanced cancer patients with uncontrolled symptoms. This is a 4-week treatment period study followed by an open label period of 1 year.

DETAILED DESCRIPTION:
This is a 4-week randomized, double-blind, placebo-controlled, parallel group design trial to evaluate the safety and efficacy of inhaled PPP001 on uncontrolled cancer pain in patients with symptoms related to advanced incurable cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent,
2. Adult male and female patients at least 18 years of age,
3. Subject agreed to follow the protocol,
4. Advanced cancer for which there is no known curative therapy as per investigator's judgement,
5. Patients experiencing at least 2 symptoms related to cancer > 4 on ESAS-r-CS NRS including pain symptom,
6. Life expectancy six weeks or longer with PPS > 50% and PaP Score Group A (30-day survival probability >70%),
7. No cognitive impairment according to Mini-Cog©,
8. The patient is able to perform deep inhalations with FEV1 more than 60%,
9. Ability to read and respond to questions in English,
10. A female volunteer must meet one of the following criteria:

    If of childbearing potential - agrees to use one of the accepted contraceptive regimens from at least 28 days prior to the first drug administration, during the study and for at least 60 days after the last dose, If of non-childbearing potential - should be surgically sterile or in a menopausal state,
11. A male volunteer with sexual partners who are pregnant, possibly pregnant, or who could become pregnant must be surgically sterile or agrees to use one of the accepted contraceptive regimens from first drug administration until 3 months after the last drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2020-07-30 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Uncontrolled cancer pain will be measured using a patient self-administered questionnaire. | change from baseline in the EORTC-QLQ-C15-PAL pain multi-item scale score at Week 4.
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 15 Palliative (EORTC-QLQ-C15-PAL). items are rated on a scale of 1 (not at all) to 4 (very much). high scores on a symptom scale correlate to increased symptom burden

SECONDARY OUTCOMES:
The overall HRQoL (Health related Quality of Life) of patients with uncontrolled symptoms related to advanced cancer will be measured using a patient self rating questionnaire. | change from baseline in the EORTC-QLQ-C15-PAL overall QoL single-item scale score at Week 4
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 15 Palliative (EORTC-QLQ-C15-PAL). single-item scale is rated from 1 (very poor) to 7 (excellent). High scores on a functional scale correspond to better functioning
The physical, emotional, and total symptom distress will be measured using a patient self administered questionnaire. | Change from Baseline in ESAS-r-CS at Weeks 1 and 4
  Revised Edmonton Symptom Assessment System (ESAS-r-CS). 11 core symptoms: pain, tiredness, nausea, depression, anxious, drowsiness, appetite, feeling of well-being, shortness of breath, constipation and trouble sleeping. 11-point NRS ranging from 0 (no symptom) to 10 (worst possible).
The palliative performance scale will be scored by a healthcare profesional. | Change from Baseline in PPS at Weeks 1 and 4
  palliative performance scale version 2 (PPSv2) for measuring functional status in end-of-life patients. A healthcare professional scores each dimension by assigning a value from 100% to 0% (death), with 10% denoting the lowest level of functioning
The satisfaction of family caregivers of patients with advanced cancer will be measured using a caregiver self administered questionnaire. | Change from Baseline in treatment-satisfaction questionnaire at Weeks 1 and 4
  The treatment satisfaction questionnaire (change version) will be used. Scale range is a left to right 7-item scale for caregiver. each item is scored from 5 (Much more satisfied now) to 1 (Much Less satisfied now).
The distress of patients with advanced cancer will be measured using a patient self-administered questionnaire | Change from Baseline in distress thermometer at Week 4
  distress thermometer adopted as a screening measure to identify and address psychological distress in individuals with cancer. Results support a cut-off score of 3 on the DT to indicate patients with clinically elevated levels of distress .

CONTACTS AND LOCATIONS:
Locations (1):
- Scottsdale Research Institute, Cave Creek, Arizona, United States

IPD SHARING:
Plan to Share IPD: No